CLINICAL TRIAL: NCT04843514
Title: Therapeutic Drug Monitoring of Asparaginase in Patients Treated on the NOPHO ALL2008 Protocol
Brief Title: TDM of Asparaginase in ALL2008
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Klug Albertsen, M.D., PhD, Associate Professor, Aarhus University Hospital
Other Study IDs: NOPHO-ALL2008-phamacokinetics
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Asparaginase is a cornerstone in the treatment of ALL. In most contemporary protocols like in NOPHO ALL2008 prolonged asparaginase treatment has been implemented.

Publish data from NOPHO ALL2008 show sufficient treatment of the majority of patients (analysing trough levels of asparaginase after 2 weeks) but 13% of the patients experience an allergic reaction to this foreign protein (85% of them after the 2nd or 3rd dose) and they have no enzyme activity even before the reaction, meaning that they don't benefit from the treatment at all. In addition 4-5% of the patients have no enzyme activity through the whole treatment without hypersensitivity symptoms. So in reality approximately 20% of the patients don't receive any asparaginase treatment. Therapeutic Drug Monitoring (TDM) of asparaginase has been established in Aarhus, Denmark, under the leadership of Birgitte Klug Albertsen (BKA). From February 2017 the centers have been invited to send samples (extended sampling) in order to gain more knowledge about the pharmacokinetics, to identify patients without activity and to establish the logistics for TDM of asparaginase, which will be mandatory in the next protocol ALLTogether, presumably opening in 2018.

From February 2016 an extended sampling for enzyme activity measurements was started and will continue until NOPHO ALL2008 closes. These samples will make it possible to do more in depth pharmacokinetic studies as well as identify the optimal sampling time points for identifying no-activity patients in the future.

A database is being developed for TDM in ALLTogether, but it will also include all the asparaginase measurements in ALL2008.

ELIGIBILITY:
Inclusion Criteria:

* ALL treated on the NOPHO ALL2008 protocol, age 1-45 years.

Exclusion Criteria:

* No samples sent

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Alle patients in the NOPHO countries aged 1-45 years treated for ALL on the NOPHO ALL2008 protocol and have asparaginase-activity-samples sent to Aarhus.
Sampling Method: Probability Sample
Enrollment: 765 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Description of the pharmacokinetics after administration of PEG-asparaginase 1000 IU/m2 in NOPHO ALL2008, cohort February 2017 and on | 2018-2021

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Denmark, Aarhus N
  - Aarhus University Hospital, Aarhus N

IPD SHARING:
Plan to Share IPD: Undecided